CLINICAL TRIAL: NCT02632344
Title: Pembrolizumab for HPV-associated Recurrent Respiratory Papilloma Patients With Laryngeal, Tracheal and/or Pulmonary Involvement
Brief Title: Pembrolizumab for HPV-associated Recurrent Respiratory Papilloma Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sara Pai, MD, PhD, Sara Pai, MD, PhD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-469
Record Dates: First submitted 2015-12-10; First posted 2015-12-16 (Estimated); Results first posted 2023-07-03 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Respiratory Papillomatosis
Keywords: Laryngeal papilloma, recurrent; Respiratory papillomatosis; Juvenile-onset recurrent respiratory papillomatosis; Human papillomavirus; Virally-related diseases
MeSH Terms: conditions — Recurrent respiratory papillomatosis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks. Treatment will be administered on Day 1 of each cycle after all procedures/assessments have been completed
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg will be administered as a 30 minute IV infusion every 3 weeks on day 1 of each cycle after all procedures/assessments have been completed.
  Other Names: Keytruda; MK-3475

SUMMARY:
This research study is evaluating an immune modulatory agent as a possible treatment for patients with Recurrent Respiratory Papillomatosis (RRP) with significant disease involving the larynx, trachea, and/or lungs. The investigators will be using Pembrolizumab as the treating agent.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. The FDA (the U.S. Food and Drug Administration) has not approved Pembrolizumab for your specific disease but it has been approved for other uses.

Pembrolizumab is a humanized monoclonal antibody. Pembrolizumab is being studied in several other clinical trials to see if it has an effect in helping the immune system to recognize and eliminate abnormal cells in the body. The antibody blocks a receptor expressed on immune cells, called T cells, and by blocking this receptor it has the potential to activate the T cells to kill abnormal cells, such as virally infected cells.

In this research study, the investigators are looking at whether Pembrolizumab can restore the natural ability of the immune system to recognize and eliminate Human papillomavirus (HPV)-infected cells from the body.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Be 12 years of age on day of signing informed consent.
* Have histologically confirmed diagnosis of RRP that involves the trachea, lungs, and/or larynx. The latter of which has required 3 or more surgeries within a year to remove the lesions from their larynx. Subjects must have evaluable disease either based on RECIST 1.1 and/or endoscopic parameters, as discussed above.
* Be required to provide tissue from a newly obtained biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to study registration. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from PI.
* Have confirmed human papillomavirus-associated lesions based on in-situ hybridization testing and/or polymerase chain reaction which may be performed on a newly obtained biopsy or archived sample.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of study registration System Laboratory Value

  * Hematological

    * Absolute neutrophil count (ANC) ≥1,500 /mcL
    * Platelets ≥100,000 / mcL
    * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
  * Renal

    * Serum creatinine OR Measured or calculated creatinine clearance ≤1.5 X upper limit of normal (ULN) OR
    * (GFR can also be used in place of creatinine or CrCl) ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
  * Hepatic

    * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
    * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
    * Albumin >2.5 mg/dL
  * Coagulation

    * International Normalized Ratio (INR) or Prothrombin Time (PT)≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
    * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
  * Creatinine clearance should be calculated per institutional standard.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving any dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. The methods of surgical sterilization include having had a hysterectomy (removal of the uterus), bilateral oophorectomy (removal of both ovaries), tubal ligation (having your tubes tied), and transvaginal occlusion (blocking the tubes with a coil).
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to study registration.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study registration or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study registration or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  --Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* Recovery from effects of any major surgery or significant traumatic injury at least 28 days before the first dose of study treatment. Endoscopic debridement of RRP lesions is NOT considered a major surgery
* No known diagnosis of invasive squamous cell carcinoma within the previous 2 years.
* Patients with invasive squamous cell carcinoma derived from their RRP who are not considered appropriate for surgery, radiation therapy, or chemotherapy by their treating oncology team may be considered eligible for the study.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. --Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04; Primary Completion 2022-02 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Pai, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - NorthShore University HealthSystem, Evanston, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 21
Completed | 13
Not Completed | 8
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab: Pembrolizumab 200 mg every 3 weeks.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 45 [19 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 2
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Via Endoscopic Lesional Burden Score and/or RECIST
Description: A Simon two-stage design was used to assess best objective response rate based on endoscopic lesional burden and Response Evaluation Criteria in Solid Tumors (RECIST). For the endoscopic lesions burden score,T=the range of the score is 0 to 83. A lower score means decreased disease burden.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 21
Participants | 21

2. Primary Outcome: Number of Participants With Adverse Events Through CTCAE
Description: To determine the safety and tolerability of pembrolizumab in subjects with RRP.
Time Frame: Up to 3 years after enrollment of the last the patient
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 21
Participants | 15

3. Secondary Outcome: Assess Duration of Response
Description: To evaluate the response duration in subjects receiving pembrolizumab.
Time Frame: Time from observed partial response to the development of progressive disease.
Population: Duration of Response was assessed among those participants who achieved a partial response (PR).
Measure: Mean (Standard Deviation); unit: months
Groups:
- Pembrolizumab: Pembrolizumab 200 mg was administered as a 30 minute IV infusion every 3 weeks on day 1 of each cycle after all procedures/assessments have been completed.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 11
months | 13.1 (6.2)

ADVERSE EVENTS:
Time Frame: Up to 3 years after study registration.
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 3/21
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=21)
Hypophysitis (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=21)
Fatigue (General disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT02632344/Prot_SAP_000.pdf